CLINICAL TRIAL: NCT02041585
Title: The Contribution of Low Physical Function, Emotional Function and Social Support to Rehospitalization Risk Among Older Adults
Brief Title: Discharge Functional Status and Rehospitalization in the Elderly
Acronym: DC PROMIS
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Luke Hansen, Assistant Professor, Northwestern University
Other Study IDs: DCPROMIS
Record Dates: First submitted 2014-01-15; First posted 2014-01-22 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Social Isolation; Depression; Anxiety; Debility
Keywords: Hospital Readmission; Social Isolation and Hospital Readmission; Age and Hospital Readmission; Functional Status and Hospital Readmission; Charlson Score and Hospital Readmission; Length of Stay and Hospital Readmission
MeSH Terms: conditions — Social Isolation; Depression; Anxiety Disorders; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elder discharge cohort: There will be no intervention in this observational survey research.

SUMMARY:
The DC PROMIS Study (also known as the Discharge Patient Reported Outcomes Measurement Information System Study) is a study to see the effect of patients' social, physical and mental function on their health after hospital discharge.

DETAILED DESCRIPTION:
Background:

Rehospitalization within 30 days of discharge is observed in approximately 19% of Medicare Fee for Service patients following discharge. Risk factors including medical comorbidity and discharge process quality have been identified as contributing to this outcome, however the possibility that patient level social and functional characteristics has not been equally investigated.

Procedural summary:

Patients will be recruited at the time of discharge. Participation in the study will include three surveys (one at the time of discharge, one within 72-96 hours after discharge and one thirty days after discharge) about functional status. The survey will inquire about function in six domains: physical function, depression, anxiety, cognition, social isolation, instrumental social support. The initial survey will be conducted in person at the hospital bedside by a research team member. The second and third surveys will be conducted by telephone within 72 to 96 day hours of discharge. Survey responses will be collected by direct patient response into tablet computer hardware.

Recruitment:

The research team (PI or RA) will identify candidates for recruitment based on conversation with the hospital case management staff and hospitalist physicians at the time of daily interdisciplinary care rounds. Inclusion criteria are age greater than or equal to 65 and anticipated return to home-based care at discharge or within two weeks of discharge. Exclusion criteria are non-English speaking language status, inability to complete interview based on sensory limitations, Mini-Cog evaluation consistent with dementia, or physician caregiver recommendation that patient not be enrolled.

Risk:

Participation in this study will not involve any physical risk beyond that of every day life. Risk will be minimized as no invasive interventions will be used. The possibility of psychological stress exists as individuals participate in interviews and complete survey items designed to test performance. Subjects may feel embarrassed to report areas of functional limitation.

Risk of emotional harm will be minimized through the supportive presence of the PI and/or RA at the time of data collection and the use of geriatric appropriate strategies for interviewing. The patient will only be approached with hospital physician recommendation.

Data Safety Primary data will be de-identified and carefully maintained in a locked area.

ELIGIBILITY:
Inclusion Criteria:

* patients cared for on the inpatient general medical and surgical services at Northwestern Memorial Hospital (NMH)
* age upon admission ≥65 years
* anticipated disposition to home at discharge or within two weeks of discharge

Exclusion Criteria:

* previous hospitalization within 30 days
* in-hospital death
* transfer to another inpatient facility at the time of discharge
* non-English language fluency
* hospital medicine attending attestation that patient is not competent or clinically stable to participate
* Mini-cog evaluation consistent with dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: General medical service inpatient hospitalist service population, aged greater than or equal to 65
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
30 day rehospitalization | Measured at 30 days following hospital discharge
  Rehospitalization is an important clinical quality/healthcare utilization measure. In this study it will be measured using patient report of rehospitalization collected via telephone followup.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Hansen, MD, MHS, Principal Investigator — Northwestern Memorial Hospital
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States